CLINICAL TRIAL: NCT03094351
Title: Robot-assisted Esophagectomy Versus Conventional Thoracoscopic Esophagectomy for Patients With Squamous Cell Esophageal Cancer: a Multicenter Open-label, Randomized Controlled Trial (RAMIE Trial)
Brief Title: Robot-assisted Esophagectomy Versus Conventional Thoracoscopic Esophagectomy
Acronym: RAE vs CTE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Ruijin Hospital (Other); Changhai Hospital (Other); Shanghai Zhongshan Hospital (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Zhigang Li, Chief, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAE20170320
Record Dates: First submitted 2017-03-20; First posted 2017-03-29 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-02

CONDITIONS: Esophageal Cancer; Esophageal Carcinoma
Keywords: robot assisted esophagectomy; minimally invasive esophagectomy; esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot assisted esophagectomy (Experimental): Robot-assisted esophagectomy with gastric conduit formation.
  Interventions: Procedure: esophagectomy
- Thoracoscopic esophagectomy (Active Comparator): Conventional thoracoscopic esophagectomy with gastric conduit formation.
  Interventions: Procedure: esophagectomy

INTERVENTIONS:
Procedure: esophagectomy — Robot assisted esophagectomy with extended two field lymphadenectomy.
  Other Names: minimally invasive esophagectomy
  Arms: Robot assisted esophagectomy
Procedure: esophagectomy — Conventional thoracoscopic esophagectomy with extended two field lymphadenectomy.
  Other Names: minimally invasive esophagectomy
  Arms: Thoracoscopic esophagectomy

SUMMARY:
This is the first randomized controlled study to compare the robot-assisted esophagectomy (RAE) to minimally invasive conventional thoracoscopic esophagectomy (CTE). The aim of this trial is to evaluate the safety, risks of the robot-assisted esophagectomy, and to compare the short-term operative outcomes and long-term oncological outcomes between the two surgical treatments.

DETAILED DESCRIPTION:
Objective: This study aims to compare the oncological outcomes between robot-assisted esophagectomy and minimally invasive conventional thoracoscopic esophagectomy.

Study design: Randomized controlled parallel-group superiority trial Study population: Patients (age >= 18 and <= 75 years) with histologically proven surgically resectable (cT1b-3, N0-2, M0) squamous cell carcinoma of the intrathoracic esophagus with European Clinical Oncology Group performance status 0, 1 or 2.

Intervention: 360 patients will be randomly allocated to either A) robot-assisted esophagectomy (n=180) or B) conventional thoracoscopic esophagectomy (n=180).

Patients will receive the following interventions:

Group A. robot assisted esophagectomy, with gastric conduit formation. Group B. conventional thoracoscopic esophagectomy, with gastric conduit formation.

Main study parameters/endpoints: Primary outcome is 5-year overall survival rate.

Secondary outcomes are 5-year disease free survival, 3-year overall survival rate, 3-year disease free survival, (in hospital) mortality within 30 and 60 days, R0 resections, operation related events, postoperative recovery, lymph nodes status, quality of life.

Follow-up: 60 months after discharge of the last randomized patient.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the intrathoracic esophagus.
* Surgical resectable (T1b-3, N0-2, M0)
* Age ≥ 18 and ≤ 75 years
* European Clinical Oncology Group performance status 0, 1 or 2
* Written informed consent

Exclusion Criteria:

* Carcinoma of the cervical esophagus
* Histologically proven adenocarcinoma or undifferentiated carcinoma.
* Prior thoracic surgery at the right hemithorax or thorax trauma.
* Infectious disease with systemic therapy indicated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2017-07-29 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival Rate | 5 years

SECONDARY OUTCOMES:
R0 resection (%) | within 30 days after surgery
Overall Survival Rate | 3 years
Disease Free Survival Rate | 3 years
Postoperative major complications | 30 days after surgery
In hospital mortality | 30-60 days after surgery
  For all patients, the cause of death will be noted. If applicable, the results of the autopsy report will be noted.
Operative duration | during the operation, up to 5 hours
  The operation time is defined as time from incision until closure (minutes) for both the thoracic phase and the abdominal phase of the procedure. For the robotic procedure, the set-up time will be recorded separately.
Postoperative recovery | from the date of surgery to the hospital discharge, assessed up to 15 days
  Postoperative hospital stay, intensive care unit (ICU) stay
Number of lymph nodes dissected | within 30 days after surgery
Quality of life | 2 years
  The quality of life assessment was based on a previously validated questionnaire, QLQ-C30 (version 3.0; quality-of-life questionnaire), combined with an esophageal cancer-specific module, QLQ-OES18.
Estimated blood loss | during the operation, up to 5 hours
Disease Free Survival Rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang Li, Master, Principal Investigator — Shanghai Chest Hospital of Shanghai Jiao Tong University; Hecheng Li, Master, Study Director — Ruijin Hospital; Hezhong Chen, Master, Study Director — Changhai Hospital, the Second Military Medical University; Lijie Tan, Master, Study Director — Fudan University; Bentong Yu, Master, Study Director — The First of Affiliated Hospital of Nanchang University
Locations (6):
- China (6):
  - General hospital of eastern theater command, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Changhai Hospital, The Second Military Medical University, Shanghai
  - Ruijin Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai
  - Shanghai Chest Hospital, Shanghai Jiao Tong University, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Y, Li B, Yi J, Hua R, Chen H, Tan L, Li H, He Y, Guo X, Sun Y, Yu B, Li Z. Robot-assisted Versus Conventional Minimally Invasive Esophagectomy for Resectable Esophageal Squamous Cell Carcinoma: Early Results of a Multicenter Randomized Controlled Trial: the RAMIE Trial. Ann Surg. 2022 Apr 1;275(4):646-653. doi: 10.1097/SLA.0000000000005023. PMID 34171870
- [Derived] Yang Y, Zhang X, Li B, Li Z, Sun Y, Mao T, Hua R, Yang Y, Guo X, He Y, Li H, Chen H, Tan L. Robot-assisted esophagectomy (RAE) versus conventional minimally invasive esophagectomy (MIE) for resectable esophageal squamous cell carcinoma: protocol for a multicenter prospective randomized controlled trial (RAMIE trial, robot-assisted minimally invasive Esophagectomy). BMC Cancer. 2019 Jun 21;19(1):608. doi: 10.1186/s12885-019-5799-6. PMID 31226960